CLINICAL TRIAL: NCT06782451
Title: Development of Preclinical Models Derived From Tumors With a Molecular Abnormality of Interest to Test Their Sensitivity to New Anti-tumor Therapies.
Acronym: DST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023/57; 2024-A01616-41 (Other: ANSM)
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-05

CONDITIONS: Neoplasm Malignant
Keywords: Spheroids; Preclinic models
MeSH Terms: conditions — Neoplasms | interventions — Surgical Procedures, Operative; Biopsy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): For this study, the included patients will have a biopsy or a surgery performed as part of routine patient care. A part of the tumor sample will be transmitted to the Laboratory of Translational Research in Oncology to develop spheroids.
  A blood sample will also be taken (38 mL) and analyzed by the Laboratory of Translational Research in Oncology in order to assess hematological toxicities of drugs and study a potential link between disease stage and the quantity of exosomes secreted.
  Interventions: Procedure: Surgery or biopsy; Procedure: Blood sample

INTERVENTIONS:
Procedure: Surgery or biopsy — A part of the tumor sample collected during the surgery or the biopsy performed as part of routine patient care will be used for the research.
Procedure: Blood sample — 38 mL of blood will be taken for the study.

SUMMARY:
This study aims to collect tumor samples from patients carrying a mutation of interest to develop a cell culture technique for "spheroids.

The goal is to use these spheroids to model responses to anticancer treatments. Various therapeutic molecules can be tested on these spheroids, enabling the evaluation of the potential of new molecules or the activity of existing ones specifically on the tumor (bearing the mutation of interest) from which the spheroid was developed.

Tumor samples will be collected as part of biopsies or surgeries conducted during routine patient care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patient for whom at least one mutation deemed of interest by the investigator has been identified.
* Patient with a malignant tumor at a locally advanced or metastatic stage, for whom a tissue tumor sample (via surgery, radiology, or endoscopy) is scheduled as part of their standard care.
* Tumor volume deemed sufficient by the physician to ensure an adequate amount of material for analysis by the pathologist and the transfer of a part of the tumor sample to the Laboratory of Translational Research in Oncology for the study.
* INR < 1.5; Platelets > 50,000/μL.
* Patient who has been informed of the study and has signed the informed consent form.
* Patient affiliated with a social security insurance.

Exclusion Criteria:

* Patient with multiple primary malignant tumors.
* Patient with a known HIV, Hepatitis C, or Hepatitis B infection.
* Patient on:

  * Clopidogrel (hydrogensulfate) or Prasugrel (hydrochloride) or Ticlopidine (hydrochloride) with no possibility of suspension for 5 days,
  * Low molecular weight heparin with no possibility of dose suspension before the procedure,
  * Fondaparinux with no possibility of suspension,
  * Abciximab with no possibility of suspension for 24 hours and aPTT < 50s and ACT < 150s,
  * Eptifibatide or Tirofiban Hydrochloride Monohydrate or Argatroban with no possibility of suspension 4 hours before the procedure,
  * Bivalirudin with no possibility of suspension 2-3 hours if CrCL >50 mL/min or 3-5 hours if CrCL <50 mL/min before the procedure,
  * Dabigatran etexilate with no possibility of suspension 2-3 days if CrCL >50 mL/min or 3-5 days if CrCL <50 mL/min before the procedure.
* Patient considered vulnerable; vulnerable persons are defined in articles L1121-5 to L1121-8:

  * Pregnant women, parturients, and breastfeeding mothers,
  * Individuals deprived of their liberty by a judicial or administrative decision, individuals hospitalized without consent under articles L. 3212-1 and L. 3213-1 who do not fall under the provisions of article L. 1121-8, and individuals admitted to a healthcare or social facility for reasons other than research,
  * Adults under legal protection or unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2030-07-02 (Estimated); Study Completion 2030-07-02 (Estimated)

PRIMARY OUTCOMES:
Development of a cell culture technique for spheroids derived from fresh tumor samples collected among patients carrying a mutation of interest. | 1 month
  The primary evaluation criterion is the percentage of patients for whom viable spheroids were obtained from tumors with a molecular abnormality of interest, measured by cell viability one month after the tumor sample was collected.

SECONDARY OUTCOMES:
Obtain spheroids that are phenotypically and genotypically stable. | 1 month
  The phenotypic and genotypic stability of spheroids over time will be assessed using molecular characterization techniques (e.g., immunohistochemistry, sequencing).
Validate preclinical models to study the tumor response to innovative therapies. | 1 month
  The ability of spheroids to mimic aspects of the tumor microenvironment, such as hypoxia and extracellular matrix formation, will be evaluated.
Test the efficacy of molecules targeting variations identified in these tumors. | 1 month
  The response of the spheroids to specific anti-tumor therapies will be evaluated through drug sensitivity tests (e.g., cytotoxicity assays).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided